CLINICAL TRIAL: NCT03857217
Title: Post-Cardiotomy Extra-Corporeal Life Support Study: a Retrospective International Multicenter Cohort Study
Brief Title: Post-Cardiotomy Extra-Corporeal Life Support Study
Acronym: PELS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL69209.068.19
Record Dates: First submitted 2019-02-19; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Cardiogenic Shock; Resuscitation; Cardiac Surgery
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Ex utero Intrapartum Treatment Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-cardiotomy patients: Patients submitted to cardiac surgery
  Interventions: Device: Extra-Corporeal Membrane Oxygenation

INTERVENTIONS:
Device: Extra-Corporeal Membrane Oxygenation — ECMO is implanted in cardiac surgery patients.

SUMMARY:
Extracorporeal life support is increasingly used after cardiac surgery. Despite improved technology, outcome still remains poor.

This retrospective multicenter cohort study aims to find the (risk) factors associated with the poor prognosis of these patients.

Adult patients who received ECLS after cardiac surgery between 2000 and 2018 are eligible for inclusion

DETAILED DESCRIPTION:
The prevalence of post-cardiotomy extracorporeal life support (PC-ECLS) reported in the literature varies between 0.6% and 3.6% of all cardiac surgical cases and has represented the most frequent indication for ECLS up to 2012.

Indications for PC-ECLS usually include intra-operative failure to wean from cardiopulmonary bypass due to perioperative left, right or biventricular failure, or refractory cardiogenic shock/cardiac arrest in the postoperative period.

Recently, The Extracorporeal Life Support Organization (ELSO) Registry reported a remarkable increase in the use of ECLS as a supportive therapy after cardiac surgery. However a disappointing trend was observed with regards to the in-hospital survival rate, reaching only 15% in the latest period.

Furthermore, despite this increase in use and new technological developments in this area, only a few comprehensive and dedicated reports about PC-ECLS have been presented. Nevertheless, PC-ECLS, has represented the main indication for ECLS utilization, and is characterized by specific aspects (duration and type of underlying disease, severity of comorbidities, indication and type of surgical procedure, modality of access and timing of implant, complication types and rates) when compared to other ECLS indications. Often these aspects are exacerbated when there is limited experience in these procedures, particularly in centers without well-established ECLS programs. All of these factors may potentially influence ECLS management and final outcomes in post-cardiotomy patients, and make this particular setting one in which there are higher risks for unfavorable results. Careful evaluation of patient features, complication rates and management, and in-hospital outcomes according to accumulated experience should provide meaningful information to assess center performance. Furthermore, analysis of overall and trends of outcomes will hopefully indicate further areas of improvement in order to improve the ECLS results. Additionally, a rather small patient cohort within the PC-ELS group, receives veno-venous (VV) support due to post-cardiotomy respiratory failure. While there is only limited data available regarding survival and predictors for a favorable outcome after post-cardiotomy VV-ECMO, these patients will be included in the current trial as well, potentially clarifying additional predictors for survival in this specific patient group. Finally, Extracorporeal carbon-dioxide removal (ECCOR) has as added a new dimension to the intensive care management of acute cardiac and/or respiratory failure in adult patient care. However, regarding post-cardiotomy patients, no studies have been published before. Therefore, as an additional subject, patients receiving ECCOR-support as an ECLS modality after cardiac surgery will be included to the current study as well in order to provide the first post-cardiotomy ECCOR results.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery prior to Extracorporeal Life Support (ECLS: VA-ECMO, VV-ECMO, ECCOR2) / Extracorporeal Membrane Oxygenation (ECMO);
* Patients who received treatment (cardiac surgery AND adjuvant ECLS) between January 2000 and December 2018

Exclusion Criteria:

* Extra-corporeal life support (ECLS) in patients who had cardiac surgery procedures, but with implant not strictly related to surgery-related hospitalization;
* ECMO implant after discharge will not be considered.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that require ECLS after cardiac screened for inclusion
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
In-hospital survival | within 30 days (expected)
  to assess the rate of survival
Intra-operative death | within 30 days (expected)
  To assess the intra-operative rate of death.
Long-term death | within 1-year
  To assess the rate of death at long-term follow-up

SECONDARY OUTCOMES:
Adverse events | during the hospitalization (within 2 months: expected)
  Rethoracotomy for bleeding, Acute Renal Insufficiency, Respiratory insufficiency, Pneumonia, Adult Respiratory Distress Syndrome (ARDS), Postoperative Transient Ischemic Attack (TIA), Postoperative Stroke, Vasoplegic syndrome, Postoperative Right Ventricular Dysfunction, Leg Ischemia, Leg Fasciotomy, Gastro-Intestinal Complications, Laparotomy
Cardiac-related death | during the hospitalization (within 2 months: expected)
  Death for cardiac disease
Qualify of file | during the hospitalization (within 2 months: expected)
  To assess the change in the quality of life after the procedure. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems: Level 1: indicating no problem; Level 2: indicating slight problems; Level 3: indicating moderate problems; Level 4: indicating severe problems; Level 5: indicating extreme problems. Higher scores indicate higher levels of health. An unique health state is defined by combining 1 level from each of the 5 dimensions. A total of 3125 possible health states is defined in this way. Each state is referred to in terms of a 5 digit code. For example state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Result] Elsharkawy HA, Li L, Esa WA, Sessler DI, Bashour CA. Outcome in patients who require venoarterial extracorporeal membrane oxygenation support after cardiac surgery. J Cardiothorac Vasc Anesth. 2010 Dec;24(6):946-51. doi: 10.1053/j.jvca.2010.03.020. PMID 20599396
- [Result] Rastan AJ, Dege A, Mohr M, Doll N, Falk V, Walther T, Mohr FW. Early and late outcomes of 517 consecutive adult patients treated with extracorporeal membrane oxygenation for refractory postcardiotomy cardiogenic shock. J Thorac Cardiovasc Surg. 2010 Feb;139(2):302-11, 311.e1. doi: 10.1016/j.jtcvs.2009.10.043. PMID 20106393
- [Result] Whitman GJ. Extracorporeal membrane oxygenation for the treatment of postcardiotomy shock. J Thorac Cardiovasc Surg. 2017 Jan;153(1):95-101. doi: 10.1016/j.jtcvs.2016.08.024. Epub 2016 Aug 31. PMID 27666787
- [Result] Saxena P, Neal J, Joyce LD, Greason KL, Schaff HV, Guru P, Shi WY, Burkhart H, Li Z, Oliver WC, Pike RB, Haile DT, Schears GJ. Extracorporeal Membrane Oxygenation Support in Postcardiotomy Elderly Patients: The Mayo Clinic Experience. Ann Thorac Surg. 2015 Jun;99(6):2053-60. doi: 10.1016/j.athoracsur.2014.11.075. Epub 2015 Apr 10. PMID 25865760
- [Result] Fukuhara S, Takeda K, Garan AR, Kurlansky P, Hastie J, Naka Y, Takayama H. Contemporary mechanical circulatory support therapy for postcardiotomy shock. Gen Thorac Cardiovasc Surg. 2016 Apr;64(4):183-91. doi: 10.1007/s11748-016-0625-4. Epub 2016 Feb 13. PMID 26874519
- [Result] Sauer CM, Yuh DD, Bonde P. Extracorporeal membrane oxygenation use has increased by 433% in adults in the United States from 2006 to 2011. ASAIO J. 2015 Jan-Feb;61(1):31-6. doi: 10.1097/MAT.0000000000000160. PMID 25303799
- [Result] McCarthy FH, McDermott KM, Kini V, Gutsche JT, Wald JW, Xie D, Szeto WY, Bermudez CA, Atluri P, Acker MA, Desai ND. Trends in U.S. Extracorporeal Membrane Oxygenation Use and Outcomes: 2002-2012. Semin Thorac Cardiovasc Surg. 2015 Summer;27(2):81-8. doi: 10.1053/j.semtcvs.2015.07.005. Epub 2015 Jul 22. PMID 26686427
- [Result] Song JH, Woo WK, Song SH, Kim HH, Kim BJ, Kim HE, Kim do J, Suh JW, Shin YR, Park HK, Lee SH, Joo HC, Lee S, Chang BC, Yoo KJ, Kim YS, Youn YN. Outcome of veno-venous extracorporeal membrane oxygenation use in acute respiratory distress syndrome after cardiac surgery with cardiopulmonary bypass. J Thorac Dis. 2016 Jul;8(7):1804-13. doi: 10.21037/jtd.2016.05.86. PMID 27499972
- [Result] Nakamura H, Yamaguchi H, Amano A, Nakao T. Venovenous extracorporeal membrane oxygenation is effective against post-cardiotomy acute respiratory failure in adults. Gen Thorac Cardiovasc Surg. 2013 Jul;61(7):402-8. doi: 10.1007/s11748-013-0226-4. Epub 2013 Feb 24. PMID 23436039
- [Result] Shekar K, Mullany DV, Thomson B, Ziegenfuss M, Platts DG, Fraser JF. Extracorporeal life support devices and strategies for management of acute cardiorespiratory failure in adult patients: a comprehensive review. Crit Care. 2014 May 9;18(3):219. doi: 10.1186/cc13865. PMID 25032748
- [Derived] Bunge JJH, Mariani S, Meuwese C, van Bussel BCT, Di Mauro M, Wiedeman D, Saeed D, Pozzi M, Loforte A, Boeken U, Samalavicius R, Bounader K, Hou X, Buscher H, Salazar L, Meyns B, Herr D, Matteucci S, Sponga S, MacLaren G, Russo C, Formica F, Sakiyalak P, Fiore A, Camboni D, Raffa GM, Diaz R, Wang IW, Jung JS, Belohlavek J, Pellegrino V, Bianchi G, Pettinari M, Barbone A, Garcia JP, Shekar K, Whitman GJR, Gommers D, Dos Reis Miranda D, Lorusso R; Post-Cardiotomy Extracorporeal Life Support (PELS-1) Investigators. Characteristics and Outcomes of Prolonged Venoarterial Extracorporeal Membrane Oxygenation After Cardiac Surgery: The Post-Cardiotomy Extracorporeal Life Support (PELS-1) Cohort Study. Crit Care Med. 2024 Oct 1;52(10):e490-e502. doi: 10.1097/CCM.0000000000006349. Epub 2024 Jun 7. PMID 38856631
- [Derived] Mariani S, Heuts S, van Bussel BCT, Di Mauro M, Wiedemann D, Saeed D, Pozzi M, Loforte A, Boeken U, Samalavicius R, Bounader K, Hou X, Bunge JJH, Buscher H, Salazar L, Meyns B, Herr D, Matteucci MLS, Sponga S, MacLaren G, Russo C, Formica F, Sakiyalak P, Fiore A, Camboni D, Raffa GM, Diaz R, Wang IW, Jung JS, Belohlavek J, Pellegrino V, Bianchi G, Pettinari M, Barbone A, Garcia JP, Shekar K, Whitman GJR, Lorusso R; PELS-1 Investigators *. Patient and Management Variables Associated With Survival After Postcardiotomy Extracorporeal Membrane Oxygenation in Adults: The PELS-1 Multicenter Cohort Study. J Am Heart Assoc. 2023 Jul 18;12(14):e029609. doi: 10.1161/JAHA.123.029609. Epub 2023 Jul 8. PMID 37421269